CLINICAL TRIAL: NCT00475033
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in Canada
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-3008
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Results first posted 2010-06-04 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Vaccines, Pneumococcal Conjugate Vaccine
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- 2 (Active Comparator)
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — 13-valent pneumococcal conjugate vaccine administered at 2-, 4-, 6-, and 12 months of age.
  Arms: 1
Biological: 7-valent pneumococcal conjugate vaccine — 7-valent pneumococcal conjugate vaccine administered at 2-, 4-, 6-, and 12 months of age.
  Arms: 2

SUMMARY:
The purpose of this study will be to evaluate the safety, tolerability and immunogenicity of 13-valent pneumococcal conjugate vaccine in healthy infants given with routine pediatric vaccinations in Canada. Immune responses induced by the infant series (NeisVac-C® and Pentacel®)and toddler dose(NeisVac-C®)of routine pediatric vaccines when administered with 13-valent pneumococcal conjugate vaccine will be studied for noninferiority to the immune responses when administered with 7-valent pneumococcal conjugate vaccine. Safety profile and immunogenicity of 13-valent pneumococcal conjugate vaccine will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month old infants (42 to 98 days)
* Available for the duration of the study and reachable by telephone

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal, Hib conjugate, diphtheria, tetanus, pertussis, polio, or meningococcal vaccine
* Previous anaphylactic reaction to any vaccine or vaccine-related component.
* Bleeding disorder, immune deficiency or suppression, or significant chronic or congenital disease
* Receipt of blood products or gamma globulin

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 603 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Canada, clintrialparticipation@wyeth.com
Locations (9):
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Coquitlam, British Columbia
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Montreal, Quebec
  - Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Canada from June 2007 through November 2007.
Groups:
- 13vPnC: Subjects received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose), co-administered with Pentacel® (a commercially available combination diphtheria, tetanus, acellular pertussis, inactivated polio and Haemophilus influenzae type b [Hib] conjugate vaccine ) at 2, 4, and 6 months of age; NeisVac-C® (a commercially available meningococcal C tetanus toxoid conjugate vaccine) at 2 and 6 months of age (infant series) and 12 months of age (toddler dose); a single type of commercially available Measles, Mumps, and Rubella vaccine (MMR) at 12 months; and a single type of commercially available varicella vaccine at 12 months of age.
- 7vPnC: Subjects received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose), co-administered with Pentacel® (a commercially available combination diphtheria, tetanus, acellular pertussis, inactivated polio and Hib conjugate vaccine ) at 2, 4, and 6 months of age; NeisVac-C® (a commercially available meningococcal C tetanus toxoid conjugate vaccine) at 2 and 6 months of age (infant series) and 12 months of age (toddler dose); a single type of commercially available MMR at 12 months; and a single type of commercially available varicella vaccine at 12 months of age.
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 300 | 303
Vaccinated Dose 1 | 300 | 303
Vaccinated Dose 2 | 297 | 296
Vaccinated Dose 3 | 293 | 294
Completed | 293 | 290
Not Completed | 7 | 13
Not completed — Failed to return | 3 | 4
Not completed — Parent or legal guardian request | 1 | 5
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 0 | 2
Period: After the Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 293 | 290
Withdrawn After Infant Series | 6 | 8
Completed | 287 | 282
Not Completed | 6 | 8
Not completed — Adverse Event | 0 | 4
Not completed — Parent or legal guardian request | 2 | 2
Not completed — Failed to return | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 0 | 1
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 287 (Vaccinated Toddler Dose) | 282 (Vaccinated Toddler Dose)
Completed | 283 | 282
Not Completed | 4 | 0
Not completed — Parent or legal guardian request | 2 | 0
Not completed — Failed to return | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 300 | 303 | 603
Age Continuous [Mean (Standard Deviation); unit: months] — Age at enrollment
  months | 2.1 (0.3) | 2.1 (0.3) | 2.1 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 152 | 295
  Male | 157 | 151 | 308

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Predefined Antibody Level ≥1:8 for Meningococcal C Serum Bactericidal Assay (SBA) in the 13vPnC Group Relative to 7vPnC Group After 2 Doses of NeisVac-C® in the Infant Series
Description: Percentage of subjects achieving predefined antibody threshold ≥1:8 along with the corresponding 95 percent (%) confidence interval (CI) for concomitant antigen meningococcal C SBA are presented. Non-inferiority was declared if the lower limit of the 2-sided 95% CI for the difference between the 2 treatment groups > -10%.
Time Frame: 1 month after 2 doses of NeisVac-C® in the infant series (7 months of age)
Population: Evaluable immunogenicity population: had treatments as randomized at all expected doses, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations. N=number of participants analyzed with a determinate post-infant series antibody concentration to the given antigen.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 284 | 278
percentage of subjects | 96.8 [94.1 to 98.5] | 99.3 [97.4 to 99.9]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Meningococcal C: Difference in proportions (13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided 95% CI for the difference between the 2 treatment groups was > -10%; Difference = -2.4, 95% CI 2-sided [-5.3 to -0.1] — Exact 2-sided CI for the difference in proportions (13vPnC, 7vPnC) expressed as a percentage

2. Primary Outcome: Geometric Mean Titer (GMT) of Meningococcal C Antigen in the 13vPnC Group Relative to 7vPnC Group After 2 Doses of NeisVac-C® in the Infant Series
Description: Antibody geometric mean titer of meningococcal C antigen are presented. GMT and corresponding 2-sided 95% CI were constructed by back transformation of the CI for the mean of the logarithmically transformed assay results computed using the Student t distribution. In addition, the 2-sided 95% confidence interval on the ratio of the geometric means for 13vPnC relative to 7vPnC was constructed by back transformation of the Student t distribution for the mean difference of the measures on the logarithmic scale.
Time Frame: 1 month after 2 doses of NeisVac-C® in the infant series (7 months of age)
Population: The evaluable immunogenicity population was the primary analysis population; N=number of participants analyzed with a determinate antibody titer to the given antigen. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 284 | 278
GMT | 361.16 [305.46 to 427.00] | 302.55 [263.89 to 346.86]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Ratio of GMs (13vPnC, 7vPnC); Test type: Superiority or Other; Ratio of geometric means = 1.19, 95% CI 2-sided [0.96 to 1.48] — CI for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC, 7vPnC)

3. Primary Outcome: Percentage of Subjects Achieving Predefined Antibody Level to Pertussis Antigens in the 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series
Description: Percentage of subjects achieving predefined antibody threshold ≥5 enzyme-linked immunosorbent assay (ELISA) units per mL (EU/mL) along with the corresponding 95 % CI for concomitant antigens pertussis (pertussis toxoid [PT], filamentous hemagglutinin [FHA], and pertactin [PRN]) and ≥ 2.2 EU/mL fimbrial agglutinogens (FIM) are presented. Non-inferiority was declared if the lower limit of the 2-sided 95% CI for the difference between the 2 treatment groups > -10%.
Time Frame: 1 month after the 3-dose infant series (7 months of age)
Population: The evaluable immunogenicity population was the primary analysis population; (n)=number of participants with an antibody concentration (titer) ≥ to prespecified level for the given antigen for 13vPnC and 7vPnC, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 300 | 303
percentage of subjects
  PT ≥5 EU/mL (n=282, 277) | 99.6 [98.0 to 100.0] | 99.6 [98.0 to 100.0]
  FHA ≥5 EU/mL (n=283, 278) | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0]
  PRN ≥5 EU/mL (n=283, 277) | 97.9 [95.4 to 99.2] | 96.8 [93.9 to 98.5]
  FIM ≥2.2 EU/mL (n=282, 275) | 95.4 [92.2 to 97.5] | 97.5 [94.8 to 99.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; PT: Difference in proportions (13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI 2-sided [-1.6 to 1.7] — Exact 2-sided CI for the difference in proportions (13vPnC, 7vPnC) expressed as a percentage
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; FHA: Difference in proportions (13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI 2-sided [-1.3 to 1.3] — Exact 2-sided CI for the difference in proportions (13vPnC, 7vPnC) expressed as a percentage
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; PRN: Difference in proportions (13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 1.1, 95% CI 2-sided [-1.7 to 4.2] — Exact 2-sided CI for the difference in proportions (13vPnC, 7vPnC) expressed as a percentage
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; FIM: Difference in proportions (13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -2.1, 95% CI 2-sided [-5.5 to 1.2] — Exact 2-sided CI for the difference in proportions (13vPnC, 7vPnC) expressed as a percentage

4. Secondary Outcome: Percentage of Subjects Achieving Predefined Antibody Level ≥1:8 for Meningococcal C SBA in the 13vPnC Group Relative to 7vPnC Group After the Toddler Dose of NeisVac-C®
Description: Percentage of subjects achieving predefined antibody threshold ≥1:8 along with the corresponding 95% CI for concomitant antigen meningococcal C SBA are presented. Non-inferiority was declared if the lower limit of the 2-sided 95% CI for the difference between the 2 treatment groups > -10%.
Time Frame: 1 month after the toddler dose of NeisVac-C® (13 months of age)
Population: The evaluable immunogenicity population was the primary analysis population. N=number of participants analyzed with a determinate post-toddler dose antibody concentration (titer) to the given antigen.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 265 | 268
percentage of subjects | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Meningococcal C: Difference in proportions (13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI 2-sided [-1.4 to 1.4] — Exact 2-sided CI for the difference in proportions (13vPnC, 7vPnC) expressed as a percentage

5. Secondary Outcome: Geometric Mean Titer (GMT) of Meningococcal C Antigen in the 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Description: Antibody geometric mean titer of meningococcal C antigen are presented. GMT and corresponding 2-sided 95% CI were constructed by back transformation of the CI for the mean of the logarithmically transformed assay results computed using the Student t distribution. In addition, the 2-sided 95% confidence interval on the ratio of the GMs for 13vPnC relative to 7vPnC was constructed by back transformation of the Student t distribution for the mean difference of the measures on the logarithmic scale.
Time Frame: 1 month after the toddler dose (13 months of age)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 265 | 268
GMT | 1379.75 [1235.06 to 1541.39] | 1083.96 [962.54 to 1220.69]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Meningococcal C: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Ratio of geometric means = 1.27, 95% CI 2-sided [1.08 to 1.50] — [estimate comment as in outcome 2, analysis 1]

6. Other Pre Specified Outcome: Percentage of Subjects Achieving Pneumococcal Immunoglobulin G (IgG) Antibody Level ≥0.35 μg/mL in the 13vPnC Group After the 3-dose Infant Series
Description: Percentage of subjects achieving World Health Organization (WHO) predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: 1 month after the 3-dose infant series (7 months of age)
Population: The evaluable immunogenicity population was the primary analysis population; (n)=number of participants with a determinate IgG antibody concentration to the given serotype for 13vPnC.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- 13vPnC: Subjects received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose). Co-administered with Pentacel® (a commercially available combination diphtheria, tetanus, acellular pertussis, inactivated polio and Haemophilus influenzae type b [Hib] conjugate vaccine ) at 2, 4, and 6 months of age; NeisVac-C® (a commercially available meningococcal C tetanus toxoid conjugate vaccine) at 2 and 6 months of age (infant series) and 12 months of age (toddler dose); a single type Measles, Mumps, and Rubella vaccine (MMR) at 12 months; and a single type of commercially available varicella vaccine at 12 months of age.
Arm/Group | 13vPnC
Number analyzed (Participants) | 300
percentage of subjects
  Common serotypes - serotype 4 (n=277) | 97.1 [94.4 to 98.7]
  Common serotypes - serotype 6B (n=276) | 93.1 [89.5 to 95.8]
  Common serotypes - serotype 9V (n=277) | 95.3 [92.1 to 97.5]
  Common serotypes - serotype 14 (n=275) | 98.2 [95.8 to 99.4]
  Common serotypes - serotype 18C n=277) | 96.4 [93.5 to 98.3]
  Common serotypes - serotype 19F (n=273) | 98.5 [96.3 to 99.6]
  Common serotypes - serotype 23F (n=275) | 90.2 [86.0 to 93.4]
  Additional serotypes - serotype 1 (n=277) | 95.7 [92.6 to 97.7]
  Additional serotypes - serotype 3 (n=275) | 79.6 [74.4 to 84.2]
  Additional serotypes - serotype 5 (n=276) | 87.0 [82.4 to 90.7]
  Additional serotypes - serotype 6A (n=276) | 96.4 [93.4 to 98.2]
  Additional serotypes - serotype 7F (n=276) | 98.6 [96.3 to 99.6]
  Additional serotypes - serotype 19A (n=272) | 97.8 [95.3 to 99.2]

7. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Pneumococcal IgG Antibody in 13vPnC Group After the 3-dose Infant Series
Description: Antibody geometric mean concentration (GMC) as measured by μg/mL for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% CI were evaluated. 2-sided 95% CI were constructed by back transformation of the CI for the mean of the logarithmically transformed assay results computed using the Student t distribution.
Time Frame: 1 month after the 3-dose infant series (7 months of age)
Population: The evaluable immunogenicity population was the primary analysis population; (n)=number of participants with a determinate antibody concentration for the given serotype for 13vPnC.
Measure: Geometric Mean (95% Confidence Interval); unit: GMC μg/mL
Arm/Group | 13vPnC
Number analyzed (Participants) | 300
GMC μg/mL
  Common serotypes - serotype 4 (n=277) | 1.46 [1.33 to 1.60]
  Common serotypes - serotype 6B (n=276) | 2.16 [1.87 to 2.49]
  Common serotypes - serotype 9V (n=277) | 1.12 [1.03 to 1.22]
  Common serotypes - serotype 14 (n=275) | 5.43 [4.86 to 6.06]
  Common serotypes - serotype 18C (n=277) | 1.37 [1.23 to 1.52]
  Common serotypes - serotype 19F (n=273) | 2.18 [1.99 to 2.39]
  Common serotypes - serotype 23F (n=275) | 1.15 [1.03 to 1.30]
  Additional serotypes - serotype 1 (n=277) | 1.82 [1.63 to 2.04]
  Additional serotypes - serotype 3 (n=275) | 0.63 [0.58 to 0.70]
  Additional serotypes - serotype 5 (n=276) | 0.90 [0.81 to 0.99]
  Additional serotypes - serotype 6A (n=276) | 1.92 [1.73 to 2.12]
  Additional serotypes - serotype 7F (n=276) | 2.26 [2.09 to 2.45]
  Additional serotypes - serotype 19A (n=272) | 2.00 [1.82 to 2.19]

8. Other Pre Specified Outcome: Percentage of Subjects Achieving Pneumococcal Immunoglobulin G (IgG) Antibody Level ≥0.35 μg/mL in the 13vPnC Group After the Toddler Dose
Description: Percentage of subjects achieving WHO predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: 1 month after the toddler dose (13 months of age)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 13vPnC
Number analyzed (Participants) | 287
percentage of subjects
  Common serotypes - serotype 4 (n=264) | 100.0 [98.6 to 100.0]
  Common serotypes - serotype 6B (n=263) | 100.0 [98.6 to 100.0]
  Common serotypes - serotype 9V (n=264) | 99.2 [97.3 to 99.9]
  Common serotypes - serotype 14 (n=264) | 100.0 [98.6 to 100.0]
  Common serotypes - serotype 18C (n=262) | 98.9 [96.7 to 99.8]
  Common serotypes - serotype 19F (n=263) | 98.1 [95.6 to 99.4]
  Common serotypes - serotype 23F (n=263) | 99.6 [97.9 to 100.0]
  Additional serotypes - serotype 1 (n=264) | 100.0 [98.6 to 100.0]
  Additional serotypes - serotype 3 (n=264) | 84.8 [79.9 to 88.9]
  Additional serotypes - serotype 5 (n=264) | 98.5 [96.2 to 99.6]
  Additional serotypes - serotype 6A (n=264) | 100.0 [98.6 to 100.0]
  Additional serotypes - serotype 7F (n=264) | 100.0 [98.6 to 100.0]
  Additional serotypes - serotype 19A (n=263) | 100.0 [98.6 to 100.0]

9. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Pneumococcal IgG Antibody in 13vPnC Group After the Toddler Dose
Description: as for outcome 7
Time Frame: 1 month after the toddler dose (13 months of age)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: GMC μg/mL
Arm/Group | 13vPnC
Number analyzed (Participants) | 287
GMC μg/mL
  Common serotypes - serotype 4 (n=264) | 2.67 [2.43 to 2.92]
  Common serotypes - serotype 6B (n=263) | 9.83 [8.83 to 10.94]
  Common serotypes - serotype 9V (n=264) | 2.04 [1.87 to 2.23]
  Common serotypes - serotype 14 (n=264) | 7.58 [6.86 to 8.37]
  Common serotypes - serotype 18C (n=262) | 2.00 [1.80 to 2.21]
  Common serotypes - serotype 19F (n=263) | 5.70 [5.06 to 6.42]
  Common serotypes - serotype 23F (n=263) | 3.59 [3.21 to 4.01]
  Additional serotypes - serotype 1 (n=264) | 3.45 [3.11 to 3.82]
  Additional serotypes - serotype 3 (n=264) | 0.74 [0.67 to 0.81]
  Additional serotypes - serotype 5 (n=264) | 2.38 [2.15 to 2.62]
  Additional serotypes - serotype 6A (n=264) | 6.47 [5.87 to 7.12]
  Additional serotypes - serotype 7F (n=264) | 3.88 [3.59 to 4.21]
  Additional serotypes - serotype 19A (n=263) | 8.36 [7.61 to 9.19]

10. Primary Outcome: Geometric Mean Concentration (GMC) of Pertussis Antigens in the 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series
Description: Antibody geometric mean concentration of pertussis antigens (PT, FHA, PRN, and FIM) as measured by EU/mL are presented. GMC and corresponding 2-sided 95% CI were constructed by back transformation of the CI for the mean of the logarithmically transformed assay results computed using the Student t distribution. In addition, the 2-sided 95% confidence intervals on the ratio of the GMCs for 13vPnC relative to 7vPnC were constructed by back transformation of the Student t distribution for the mean difference of the measures on the logarithmic scale.
Time Frame: 1 month after the 3-dose Infant Series (7 months of age)
Population: The evaluable immunogenicity population was the primary analysis population; (n)=number of participants with a determinate antibody concentration (titer) to the given antigen. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: GMC EU/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 300 | 303
GMC EU/mL
  PT (n=282, 277) | 46.06 [42.83 to 49.53] | 40.37 [37.24 to 43.75]
  FHA (n=283,278) | 78.08 [72.47 to 84.13] | 69.52 [64.39 to 75.05]
  PRN (n=283, 277) | 42.90 [38.17 to 48.22] | 40.69 [36.16 to 45.79]
  FIM (n=282, 275) | 11.54 [10.48 to 12.71] | 12.98 [11.81 to 14.27]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; PT: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Ratio of geometric means = 1.14, 95% CI 2-sided [1.02 to 1.27] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; FHA: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Ratio of geometric means = 1.12, 95% CI 2-sided [1.01 to 1.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; PRN: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Ratio of geometric means = 1.05, 95% CI 2-sided [0.89 to 1.24] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; FIM: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Ratio of geometric means = 0.89, 95% CI 2-sided [0.78 to 1.02] — [estimate comment as in outcome 2, analysis 1]

11. Primary Outcome: Percentage of Subjects Achieving Predefined Antibody Level ≥0.15 Micrograms Per mL (μg/mL) for Polyribosylribitol Phosphate (PRP) in Hib in the 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series
Description: Percentage of subjects achieving predefined antibody threshold ≥0.15 μg/mL along with the corresponding 95 percent (%) confidence interval (CI) for concomitant antigen PRP in Hib are presented. Non-inferiority was declared if the lower limit of the 2-sided 95% CI for the difference between the 2 treatment groups > -10%.
Time Frame: 1 month after the 3-dose infant series (7 months of age)
Population: The evaluable immunogenicity population was the primary analysis population. N=number of participants analyzed with a determinate post-infant series antibody concentration to the given antigen.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 272 | 266
percentage of subjects | 97.8 [95.3 to 99.2] | 99.6 [97.9 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in proportions (13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -1.8, 95% CI 2-sided [-4.4 to 0.1] — Exact 2-sided CI for the difference in proportions (13vPnC, 7vPnC) expressed as a percentage

12. Primary Outcome: Geometric Mean Concentration (GMC) of PRP in Hib in the 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series
Description: Antibody geometric mean concentration of PRP in Hib as measured by µg/mL are presented. GMC and corresponding 2-sided 95% CI were constructed by back transformation of the CI for the mean of the logarithmically transformed assay results computed using the Student t distribution. In addition, the 2-sided 95% confidence interval on the ratio of the GMCs for 13vPnC relative to 7vPnC was constructed by back transformation of the Student t distribution for the mean difference of the measures on the logarithmic scale.
Time Frame: 1 month after the 3-dose infant series (7 months of age)
Population: The evaluable immunogenicity population was the primary analysis population; N=number of participants analyzed with a determinate antibody concentration (titer) to the given antigen. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: GMC µg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 272 | 266
GMC µg/mL | 2.87 [2.48 to 3.32] | 3.14 [2.74 to 3.60]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; PRP in Hib: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Ratio of geometric means = 0.91, 95% CI 2-sided [0.75 to 1.12] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Percentage of Subjects Achieving Predefined Antibody Level ≥1.0 μg/mL for PRP in Hib in the 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series
Description: Percentage of subjects achieving predefined antibody threshold ≥1.0 μg/mL along with the corresponding 95% CI for concomitant antigen PRP in Hib are presented. Non-inferiority was declared if the lower limit of the 2-sided 95% CI for the difference between the 2 treatment groups > -10%.
Time Frame: 1 month after the 3-dose infant series (7 months of age)
Population: The evaluable immunogenicity population was the primary analysis population. N=number of participants analyzed with a determinate post-infant series antibody concentration (titer) to the given antigen.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 272 | 266
percentage of subjects | 81.6 [76.5 to 86.0] | 84.6 [79.7 to 88.7]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; PRP: Difference in proportions (13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -3.0, 95% CI 2-sided [-9.4 to 3.4] — Exact 2-sided CI for the difference in proportions (13vPnC, 7vPnC) expressed as a percentage

14. Other Pre Specified Outcome: Percentage of Subjects Reporting Pre-specified Local Reactions in the 13vPnC and 7vPnC Groups: Infant Series Dose 1 (2 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Induration and erythema were scaled as Any (induration or erythema present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Subjects may be represented in more than 1 category.
Time Frame: Within 4 days after dose (2 months of age)
Population: Safety population: all subjects who received at least 1 dose of study vaccine. N=number of subjects reporting any local reactions; (n)=number of subjects reporting yes for at least 1 day or no for all days for the 13vPnC and 7vPnC groups, respectively.
Measure: Number; unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 284 | 284
percentage of subjects
  Tenderness: Any (n=281, 283) | 44.5 | 43.8
  Tenderness: Significant (n=270, 274) | 4.4 | 4.0
  Induration: Any (n=271, 276) | 5.9 | 7.2
  Induration: Mild (n=270, 275) | 5.6 | 5.5
  Induration: Moderate (n=267, 274) | 0.7 | 2.6
  Induration: Severe (n=266, 273) | 0.0 | 0.0
  Erythema: Any (n=270, 275) | 11.1 | 14.5
  Erythema: Mild (n=270, 275) | 10.7 | 14.2
  Erythema: Moderate (n=266, 273) | 0.4 | 0.7
  Erythema: Severe (n=266, 273) | 0.0 | 0.0

15. Other Pre Specified Outcome: Percentage of Subjects Reporting Pre-specified Local Reactions in the 13vPnC and 7vPnC Groups: Infant Series Dose 2 (4 Months of Age)
Description: as for outcome 14
Time Frame: Within 4 days after dose (4 months of age)
Population: Safety population; N=number of subjects reporting any local reactions; (n)=number of subjects reporting yes for at least 1 day or no for all days for the 13vPnC and 7vPnC groups, respectively.
Measure: Number; unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 271 | 268
percentage of subjects
  Tenderness: Any (n=264, 266) | 37.5 | 32.7
  Tenderness: Significant (n=248, 252) | 3.6 | 3.6
  Induration: Any (n=251, 253) | 10.8 | 11.5
  Induration: Mild (n=251, 253) | 10.4 | 11.5
  Induration: Moderate (n=245, 252) | 0.8 | 0.4
  Induration: Severe (n=245, 252) | 0.0 | 0.0
  Erythema: Any (n=258, 257) | 18.2 | 18.3
  Erythema: Mild (n=256, 257) | 16.8 | 17.9
  Erythema: Moderate (n=247, 252) | 2.0 | 0.8
  Erythema: Severe (n=245, 252) | 0.0 | 0.0

16. Other Pre Specified Outcome: Percentage of Subjects Reporting Pre-specified Local Reactions in the 13vPnC and 7vPnC Groups: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 14
Time Frame: Within 4 days after dose (6 months of age)
Population: as for outcome 15
Measure: Number; unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 251 | 264
percentage of subjects
  Tenderness: Any (n=245, 257) | 27.3 | 28.0
  Tenderness: Significant (n=238, 244) | 3.8 | 0.8
  Induration: Any (n=243, 250) | 11.5 | 10.0
  Induration: Mild (n=243, 250) | 11.1 | 9.6
  Induration: Moderate (n=238, 244) | 0.8 | 1.2
  Induration: Severe (n=237, 244) | 0.0 | 0.0
  Erythema: Any (n=244, 253) | 16.4 | 17.8
  Erythema: Mild (n=244, 253) | 16.4 | 17.0
  Erythema: Moderate (n=237, 244) | 0.4 | 0.8
  Erythema: Severe (n=237, 244) | 0.0 | 0.0

17. Other Pre Specified Outcome: Percentage of Subjects Reporting Pre-specified Local Reactions in the 13vPnC and 7vPnC Groups: Toddler Dose (12 Months of Age)
Description: as for outcome 14
Time Frame: Within 4 days after dose (12 months of age)
Population: as for outcome 15
Measure: Number; unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 223 | 227
percentage of subjects
  Tenderness: Any (n=216, 223) | 25.0 | 28.7
  Tenderness: Significant (n=198, 210) | 2.5 | 1.0
  Induration: Any (n=198, 213) | 11.1 | 9.4
  Induration: Mild (n=198, 213) | 10.6 | 8.9
  Induration: Moderate (n=196, 210) | 1.0 | 2.4
  Induration: Severe (n=195, 210) | 0.0 | 0.0
  Erythema: Any (n=204, 216) | 19.6 | 16.7
  Erythema: Mild (n=202, 216) | 18.8 | 14.8
  Erythema: Moderate (n=197, 210) | 2.5 | 2.4
  Erythema: Severe (n=195, 210) | 0.0 | 0.0

18. Other Pre Specified Outcome: Percentage of Subjects Reporting Pre-specified Systemic Events in the 13vPnC and 7vPnC Group: Infant Series Dose 1 (2 Months of Age)
Description: Systemic events (any fever ≥38 degrees Celsius [C], decreased appetite, irritability, increased sleep, and decreased sleep were reported using an electronic diary. Subjects may be represented in more than 1 category.
Time Frame: Within 4 days after dose (2 months of age)
Population: Safety population; N=number of subjects reporting any systemic events; (n)=number of subjects reporting yes for at least 1 day or no for all days for the 13vPnC and 7vPnC groups, respectively.
Measure: Number; unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 296 | 298
percentage of subjects
  Fever ≥38 but ≤39 degrees C (n=269, 273) | 8.9 | 9.2
  Fever >39 but ≤40 degrees C (n=267, 273) | 0.7 | 0.0
  Fever >40 degrees C (n=266, 273) | 0.0 | 0.0
  Decreased appetite (n=279, 283) | 42.7 | 36.0
  Irritability (n=291, 288) | 80.8 | 83.0
  Increased sleep (n=286, 292) | 62.9 | 64.7
  Decreased sleep (n=276, 276) | 29.7 | 28.3

19. Other Pre Specified Outcome: Percentage of Subjects Reporting Pre-specified Systemic Events in the 13vPnC and 7vPnC Group: Infant Series Dose 2 (4 Months of Age)
Description: as for outcome 18
Time Frame: Within 4 days after dose (4 months of age)
Population: as for outcome 18
Measure: Number; unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 288 | 290
percentage of subjects
  Fever ≥38 but ≤39 degrees C (n=249, 255) | 8.0 | 7.5
  Fever >39 but ≤40 degrees C (n=245, 253) | 0.4 | 0.4
  Fever >40 degrees C (n=245, 252) | 0.0 | 0.0
  Decreased appetite (n=254, 262) | 28.7 | 31.3
  Irritability (n=283, 281) | 71.0 | 70.1
  Increased sleep (n=263, 275) | 54.4 | 52.4
  Decreased sleep (n=256, 261) | 25.8 | 31.0

20. Other Pre Specified Outcome: Percentage of Subjects Reporting Pre-specified Systemic Events in the 13vPnC and 7vPnC Group: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 18
Time Frame: Within 4 days after dose (6 months of age)
Population: as for outcome 18
Measure: Number; unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 275 | 277
percentage of subjects
  Fever ≥38 but ≤39 degrees C (n=237, 244) | 8.9 | 5.7
  Fever >39 but ≤40 degrees C (n=237, 244) | 0.4 | 0.8
  Fever >40 degrees C (n=237, 244) | 0.0 | 0.0
  Decreased appetite (n=249, 253) | 33.3 | 31.2
  Irritability (n=266, 270) | 68.0 | 65.9
  Increased sleep (n=255, 258) | 35.7 | 39.9
  Decreased sleep (n=251, 254) | 29.9 | 28.3

21. Other Pre Specified Outcome: Percentage of Subjects Reporting Pre-specified Systemic Events in the 13vPnC and 7vPnC Group: Toddler Dose (12 Months of Age)
Description: as for outcome 18
Time Frame: Within 4 days after dose (12 months of age)
Population: as for outcome 18
Measure: Number; unit: percentage of subjects
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 247 | 252
percentage of subjects
  Fever ≥38 but ≤39 degrees C (n=203, 213) | 13.3 | 12.2
  Fever >39 but ≤40 degrees C (n=196, 210) | 2.0 | 1.4
  Fever >40 degrees C (n=) 195, 210 | 0.0 | 0.5
  Decreased appetite (n=211, 225) | 37.0 | 34.2
  Irritability (n=240, 241) | 68.8 | 58.5
  Increased sleep (n=212, 226) | 33.5 | 33.2
  Decreased sleep (n=212, 227) | 34.0 | 33.9

ADVERSE EVENTS:
Time Frame: Baseline through 6 Month Follow-up after last study vaccination (18 Months). Local reactions and systemic events assessed within 4 days of dose: Infant Series Dose 1, 2, and 3 at 2, 4, and 6 months of age, respectively; Toddler Dose at 12 months of age.
Description: Safety population = all randomized subjects with at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Groups:
- 13vPnC Infant Series: Subjects received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 2, 4, and 6 months of age (infant series), co-administered with Pentacel® at 2, 4, and 6 months of age; NeisVac-C® at 2 and 6 months of age (infant series).
  Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=229; systematic (solicited) Any Local Reactions N=144; systematic (solicited) Any Systemic Events N=273.
- 7vPnC Infant Series: Subjects received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 2, 4, and 6 months of age (infant series), co-administered with Pentacel at 2, 4, and 6 months of age; NeisVac-C® at 2 and 6 months of age (infant series).
  Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=230; systematic (solicited) Any Local Reactions N=148; systematic (solicited) Any Systemic Events N=279.
- 13vPnC After the Infant Series: Subjects received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 2, 4, and 6 months of age (infant series), co-administered with Pentacel® at 2, 4, and 6 months of age; NeisVac-C® at 2 and 6 months of age (infant series).
- 7vPnC After the Infant Series: Subjects received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 2, 4, and 6 months of age (infant series), co-administered with Pentacel at 2, 4, and 6 months of age; NeisVac-C® at 2 and 6 months of age (infant series).
- 13vPnC Toddler Dose: Subjects received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 12 months of age (toddler dose), co-administered NeisVac-C® at 12 months of age (toddler dose); a single type of commercially available MMR at 12 months; and a single type of commercially available varicella vaccine at 12 months of age.
  Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=110; systematic (solicited) Any Local Reactions N=84; systematic (solicited) Any Systemic Events N=199.
- 7vPnC Toddler Dose: Subjects received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 12 months of age (toddler dose), co-administered with NeisVac-C® at 12 months of age (toddler dose); a single type of commercially available MMR at 12 months; and a single type of commercially available varicella vaccine at 12 months of age.
  Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=108; systematic (solicited) Any Local Reactions N=86; systematic (solicited) Any Systemic Events N=193.
- 13vPnC Toddler Dose 6-Month Follow-up: Subjects received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) at 12 months of age (toddler dose), co-administered NeisVac-C® at 12 months of age (toddler dose); a single type of commercially available MMR at 12 months; and a single type of commercially available varicella vaccine at 12 months of age.
- 7vPnC Toddler Dose 6-Month Follow-up: Subjects received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 12 months of age (toddler dose), co-administered with NeisVac-C® at 12 months of age (toddler dose); a single type of commercially available MMR at 12 months; and a single type of commercially available varicella vaccine at 12 months of age.
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC After the Infant Series | 7vPnC After the Infant Series | 13vPnC Toddler Dose | 7vPnC Toddler Dose | 13vPnC Toddler Dose 6-Month Follow-up | 7vPnC Toddler Dose 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 5/300 | 5/303 | 11/299 | 7/301 | 2/286 | 2/280 | 7/299 | 3/301
Other Adverse Events (participants affected / at risk) | 273/300 | 279/303 | 20/299 | 16/301 | 199/286 | 193/280 | 6/299 | 4/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=300) | 7vPnC Infant Series (N=303) | 13vPnC After the Infant Series (N=299) | 7vPnC After the Infant Series (N=301) | 13vPnC Toddler Dose (N=286) | 7vPnC Toddler Dose (N=280) | 13vPnC Toddler Dose 6-Month Follow-up (N=299) | 7vPnC Toddler Dose 6-Month Follow-up (N=301)
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Developmental delay (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 4 | 3 | 2 | 2 | 0 | 0 | 3 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis meningococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Physical testicle examination abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=300) | 7vPnC Infant Series (N=303) | 13vPnC After the Infant Series (N=299) | 7vPnC After the Infant Series (N=301) | 13vPnC Toddler Dose (N=286) | 7vPnC Toddler Dose (N=280) | 13vPnC Toddler Dose 6-Month Follow-up (N=299) | 7vPnC Toddler Dose 6-Month Follow-up (N=301)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 5 | 9 | 0 | 0 | 3 | 3 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 7 | 4 | 0 | 0 | 0 | 1 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 13 | 3 | 3 | 1 | 0 | 0 | 0 | 1
Dental discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 30 | 29 | 1 | 0 | 6 | 5 | 1 | 0
Faecal volume increased (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Gingival cyst (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 16 | 14 | 0 | 0 | 1 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 22 | 19 | 0 | 0 | 8 | 5 | 1 | 0
Vomiting neonatal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting projectile (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 15 | 14 | 0 | 0 | 1 | 1 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (General disorders) | 18 | 12 | 0 | 0 | 2 | 4 | 0 | 0
Malaise (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 33 | 43 | 0 | 0 | 20 | 23 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to metals (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Milk allergy (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 12 | 11 | 0 | 0 | 3 | 3 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Candida nappy rash (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Croup infectious (Infections and infestations) | 5 | 4 | 0 | 1 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 8 | 10 | 0 | 0 | 8 | 3 | 0 | 0
Eye infection (Infections and infestations) | 4 | 5 | 0 | 0 | 3 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 13 | 12 | 0 | 0 | 2 | 3 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 68 | 60 | 0 | 1 | 10 | 13 | 0 | 0
Oral candidiasis (Infections and infestations) | 7 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 5 | 9 | 0 | 1 | 9 | 6 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Roseola (Infections and infestations) | 3 | 5 | 0 | 0 | 2 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 60 | 53 | 4 | 1 | 18 | 19 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Varicella (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Viral skin infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Accidental needle stick (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Physical examination abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 0 | 0 | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head titubation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Perineal laceration (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Crying (Psychiatric disorders) | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Listless (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital labial adhesions (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 22 | 1 | 0 | 4 | 6 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 31 | 21 | 1 | 0 | 8 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 23 | 20 | 0 | 1 | 9 | 4 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 12 | 7 | 1 | 0 | 3 | 2 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 19 | 24 | 1 | 0 | 3 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 14 | 19 | 0 | 1 | 17 | 19 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin warm (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Measles (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Measles post vaccine (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Positional plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tenderness (any) (Skin and subcutaneous tissue disorders) | 125/281 | 124/283 | 0/0 | 0/0 | 54/216 | 64/223 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 99/264 | 87/266 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (any) (Skin and subcutaneous tissue disorders) | 67/245 | 72/257 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 12/270 | 11/274 | 0/0 | 0/0 | 5/198 | 2/210 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 9/248 | 9/252 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 9/238 | 2/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)
Induration (any) (Skin and subcutaneous tissue disorders) | 16/271 | 20/276 | 0/0 | 0/0 | 22/198 | 20/213 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (any)=present at site of vaccination.
Induration (any) (Skin and subcutaneous tissue disorders) | 27/251 | 29/253 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)
Induration (any) (Skin and subcutaneous tissue disorders) | 28/243 | 25/250 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (any)
Induration (mild) (Skin and subcutaneous tissue disorders) | 15/270 | 15/275 | 0/0 | 0/0 | 21/198 | 19/213 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (mild) (Skin and subcutaneous tissue disorders) | 26/251 | 29/253 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild)
Induration (mild) (Skin and subcutaneous tissue disorders) | 27/243 | 24/250 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild)
Induration (moderate) (Skin and subcutaneous tissue disorders) | 2/267 | 7/274 | 0/0 | 0/0 | 2/196 | 5/210 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (moderate) (Skin and subcutaneous tissue disorders) | 2/245 | 1/252 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (moderate) (Skin and subcutaneous tissue disorders) | 2/238 | 3/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate)
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/266 | 0/273 | 0/0 | 0/0 | 0/195 | 0/210 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/245 | 0/252 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe)
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/237 | 0/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe)
Erythema (any) (Skin and subcutaneous tissue disorders) | 30/270 | 40/275 | 0/0 | 0/0 | 40/204 | 36/216 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (any)=present at site of vaccination.
Erythema (any) (Skin and subcutaneous tissue disorders) | 47/258 | 47/257 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any)
Erythema (any) (Skin and subcutaneous tissue disorders) | 40/244 | 45/253 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (any)
Erythema (mild) (Skin and subcutaneous tissue disorders) | 29/270 | 39/275 | 0/0 | 0/0 | 38/202 | 32/216 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (mild) (Skin and subcutaneous tissue disorders) | 43/256 | 46/257 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild)
Erythema (mild) (Skin and subcutaneous tissue disorders) | 40/244 | 43/253 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (mild)
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 1/266 | 2/273 | 0/0 | 0/0 | 5/197 | 5/210 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 5/247 | 2/252 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate)
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 1/237 | 2/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (moderate)
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/266 | 0/273 | 0/0 | 0/0 | 0/195 | 0/210 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/245 | 0/252 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe)
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/237 | 0/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (severe)
Fever ≥38 degrees Celsius (C) but ≤39 degrees C (General disorders) | 24/269 | 25/273 | 0/0 | 0/0 | 27/203 | 26/213 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38 degrees Celsius C but ≤39 degrees C (General disorders) | 20/249 | 19/255 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38 degrees C but ≤39 degrees C (General disorders) | 21/237 | 14/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38 degrees C but ≤39 degrees C
Fever >39 degrees C but ≤40 degrees C (General disorders) | 2/267 | 0/273 | 0/0 | 0/0 | 4/196 | 3/210 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39 degrees C but ≤40 degrees C
Fever >39 degrees C but ≤40 degrees C (General disorders) | 1/245 | 1/253 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39 degrees C but ≤40 degrees C
Fever >39 degrees C but ≤40 degrees C (General disorders) | 1/237 | 2/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39 degrees C but ≤40 degrees C
Fever >40 degrees C (General disorders) | 0/266 | 0/273 | 0/0 | 0/0 | 0/195 | 1/210 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40 degrees C
Fever >40 degrees C (General disorders) | 0/245 | 0/252 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40 degrees C
Fever >40 degrees C (General disorders) | 0/237 | 0/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40 degrees C
Decreased appetite (General disorders) | 119/279 | 102/283 | 0/0 | 0/0 | 78/211 | 77/225 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 73/254 | 82/262 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 83/249 | 79/253 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 235/291 | 239/288 | 0/0 | 0/0 | 165/240 | 141/241 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 201/283 | 197/281 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 181/266 | 178/270 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 180/286 | 189/292 | 0/0 | 0/0 | 71/212 | 75/226 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 143/263 | 144/275 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 91/255 | 103/258 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 82/276 | 78/276 | 0/0 | 0/0 | 72/212 | 77/227 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 66/256 | 81/261 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 75/251 | 72/254 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.